CLINICAL TRIAL: NCT00182767
Title: A Phase I/II Study of BMS-247550 and Pegylated Liposomal Doxorubicin (Doxil®) in Patients With Advanced Epithelial Ovarian Cancer or Primary Peritoneal Cancer Who Have Been Previously Treated With a Platinum and a Taxane
Brief Title: Ixabepilone and Liposomal Doxorubicin in Advanced Ovarian Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00140; NCI-2009-00140 (Other: CTRP (Clinical Trial Reporting Program)); 0504007857 (Other: Montefiore Medical Center - Moses Campus); 7229 (Other: CTEP); N01CM62204 (NIH); P30CA013330 (NIH)
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Results first posted 2016-03-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2014-02

CONDITIONS: Fallopian Tube Cancer; Female Reproductive Cancer; Recurrent Breast Cancer; Recurrent Ovarian Epithelial Cancer; Stage III Ovarian Epithelial Cancer; Stage IV Breast Cancer; Stage IV Ovarian Epithelial Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Breast Neoplasms; Carcinoma, Ovarian Epithelial | interventions — ixabepilone; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (ixabepilone and doxorubicin) (Experimental): Ixabepilone IV over 3 hours and pegylated liposomal doxorubicin hydrochloride IV over 30-60 minutes on day 1.
  Interventions: Drug: ixabepilone; Drug: pegylated liposomal doxorubicin hydrochloride

INTERVENTIONS:
Drug: ixabepilone — Given IV
  Other Names: BMS-247550; epothilone B lactam; Ixempra
Drug: pegylated liposomal doxorubicin hydrochloride — Given IV
  Other Names: CAELYX; Dox-SL; DOXIL; doxorubicin hydrochloride liposome; LipoDox

SUMMARY:
This trial is studying the side effects and best dose of ixabepilone when given together with pegylated liposomal doxorubicin hydrochloride and to see how well they work in treating women with advanced ovarian epithelial, primary peritoneal cavity, or fallopian tube cancer or metastatic breast cancer. Drugs used in chemotherapy, such as ixabepilone and pegylated liposomal doxorubicin hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose and recommended phase II dose of ixabepilone when combined with pegylated doxorubicin hydrochloride (HCl) liposome (pegylated liposomal doxorubicin hydrochloride) in women with previously treated advanced ovarian epithelial, primary peritoneal cavity, or fallopian tube cancer or metastatic breast cancer.

II. To determine the safety profile of this regimen in these patients. III. To determine the clinical efficacy of this regimen in patients with platinum- and taxane-resistant advanced ovarian epithelial, primary peritoneal cavity, or fallopian tube cancer.

OUTLINE: This is a phase I, multicenter, open-label, dose-escalation study of ixabepilone followed by a phase II study.

Patients receive ixabepilone intravenously (IV) over 3 hours and pegylated liposomal doxorubicin hydrochloride IV over 30-60 minutes on day 1. Courses repeat every 21-28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of 1 of the following: advanced ovarian epithelial, primary peritoneal cavity, or fallopian tube cancer (phase I and II) or metastatic breast cancer (phase I only).
* Platinum- and taxane-resistant disease, defined as a disease-free interval of < 6 months after completion of platinum- and taxane-based chemotherapy. Disease progression during the regimen (phase II) or previously treated with >= 2 prior regimens for metastatic breast cancer, including 1 taxane-based regimen in the adjuvant or metastatic setting (phase I).
* Meets 1 of the following criteria: Previously treated with a standard course of taxane- and platinum-based chemotherapy for ovarian epithelial, primary peritoneal cavity, or fallopian tube cancer, that is platinum-refractory or -sensitive disease (phase I );
* Measurable or evaluable disease, meeting 1 of the following criteria: unidimensionally measurable lesion, known disease and CA 125 > 50 U/mL on 2 occasions >= 1 week apart or known disease and CA 27-29, CA 15-3, or CA 125 > 50 U/mL on 2 occasions >= 1 week apart (for breast cancer patients)
* ECOG 0-2 or Karnofsky 60-100%
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered.
* At least 1 week since prior chemotherapy if given on a daily or weekly schedule and recovered.
* At least 3 weeks since prior radiotherapy and recovered.
* Recovered for more than 4 weeks from all adverse events related to prior agents.
* Normal organ function including:
* Normal bilirubin
* WBC >= 3,000/mm3
* Absolute neutrophil count >= 1,500/mm3
* Platelet count >= 100,000/mm3
* AST and ALT =< 2.5 times upper limit of normal (ULN)
* Creatinine =< 1.5 times ULN or Creatinine clearance ≥ 60 mL/min

Exclusion criteria:

* No other concurrent investigational agents.
* No concurrent combination antiretroviral therapy for HIV-positive patients.
* No other concurrent anticancer therapy.
* Has received a previous chemotherapy regimen for this cancer that included drugs such as docetaxel or paclitaxel.
* Life expectancy of more than 3 months
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to Cremophor® or study drugs
* No neuropathy >= grade 2
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance.
* No other uncontrolled illness.
* No active brain metastases, including any of the following: evidence of cerebral edema by CT scan or MRI, evidence of disease progression on prior imaging studies, requirement for steroids or clinical symptoms of brain metastasis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-01; Primary Completion 2012-04 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Chuang, Principal Investigator — Montefiore Medical Center - Moses Campus
Locations (5):
- United States (5):
  - University of Connecticut, Farmington, Connecticut
  - Women's Cancer Care Associates LLC, Albany, New York
  - Weill Medical College of Cornell University, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York

REFERENCES:
- [Result] Chuang E, Wiener N, Christos P, Kessler R, Cobham M, Donovan D, Goldberg GL, Caputo T, Doyle A, Vahdat L, Sparano JA. Phase I trial of ixabepilone plus pegylated liposomal doxorubicin in patients with adenocarcinoma of breast or ovary. Ann Oncol. 2010 Oct;21(10):2075-2080. doi: 10.1093/annonc/mdq080. Epub 2010 Mar 31. PMID 20357034

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 45 patients were enrolled and treated between January 2006 and May 2011
Groups:
- Ixabepilone: 24mg/m2 and Doxil 30 mg/m2: Level 1; Ixabepilone: 32mg/m2 and Doxil 30 mg/m2: Level 2; Ixabepilone: 40mg/m2 and Doxil 30 mg/m2: Level 3: Ixabepilone IV over 3 hours and pegylated liposomal doxorubicin hydrochloride IV over 30-60 minutes on day 1.
  ixabepilone: Given IV
  pegylated liposomal doxorubicin hydrochloride: Given IV
- Ixabepilone: 13mg/m2 and Doxil 30 mg/m2: Level 4; Ixabepilone: 16mg/m2 and Doxil 30 mg/m2: Level 5: Ixabepilone IV over 3 hours on days 1, 8 and 15 and pegylated liposomal doxorubicin hydrochloride IV over 30-60 minutes on day 1.
  ixabepilone: Given IV
  pegylated liposomal doxorubicin hydrochloride: Given IV
Period: Overall Study
Arm/Group | Ixabepilone: 24mg/m2 and Doxil 30 mg/m2: Level 1 | Ixabepilone: 32mg/m2 and Doxil 30 mg/m2: Level 2 | Ixabepilone: 40mg/m2 and Doxil 30 mg/m2: Level 3 | Ixabepilone: 13mg/m2 and Doxil 30 mg/m2: Level 4 | Ixabepilone: 16mg/m2 and Doxil 30 mg/m2: Level 5
Started | 6 | 6 | 6 | 3 | 24
Completed | 6 | 6 | 6 | 3 | 24
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Ixabepilone and Doxorubicin): Ixabepilone IV over 3 hours and pegylated liposomal doxorubicin hydrochloride IV over 30-60 minutes.
  ixabepilone: Given IV
  pegylated liposomal doxorubicin hydrochloride: Given IV
Arm/Group | Treatment (Ixabepilone and Doxorubicin)
Number analyzed (Participants) | 45
Age, Continuous [Median (Full Range); unit: years] | 59 [34 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Dose-limiting Toxicity (DLT), Graded Using the National Cancer Institute (NCI) Common Toxicity Criteria (CTC) Version 4.0 (Phase I)
Description: Dose-Limiting Toxicities are assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events classification and usually encompasses all grade 3 or higher toxicities
Time Frame: 28 days
Measure: Number; unit: participants
Groups:
- Ixabepilone 24mg/m2 and Doxorubicin 30mg/m2: Level 1; Ixabepilone 32mg/m2 and Doxorubicin 30mg/m2: Level 2; Ixabepilone 40mg/m2 and Doxorubicin 30mg/m2: Level 3: Ixabepilone IV over 3 hours and pegylated liposomal doxorubicin hydrochloride IV over 30-60 minutes on day 1 every 21 days
  ixabepilone: Given IV
  pegylated liposomal doxorubicin hydrochloride: Given IV
- Ixabepilone 13mg/m2 and Doxorubicin 30mg/m2: Level 4; Ixabepilone 16mg/m2 and Doxorubicin 30mg/m2: Level 5: Ixabepilone IV over 3 hours on days 1, 8 and 15 and pegylated liposomal doxorubicin hydrochloride IV over 30-60 minutes on day 1 every 28 days
  ixabepilone: Given IV
  pegylated liposomal doxorubicin hydrochloride: Given IV
Arm/Group | Ixabepilone 24mg/m2 and Doxorubicin 30mg/m2: Level 1 | Ixabepilone 32mg/m2 and Doxorubicin 30mg/m2: Level 2 | Ixabepilone 40mg/m2 and Doxorubicin 30mg/m2: Level 3 | Ixabepilone 13mg/m2 and Doxorubicin 30mg/m2: Level 4 | Ixabepilone 16mg/m2 and Doxorubicin 30mg/m2: Level 5
Number analyzed (Participants) | 6 | 6 | 6 | 3 | 9
participants | 1 | 1 | 2 | 0 | 0

2. Secondary Outcome: Proportion of Patients Responding to Therapy (Complete Response [CR], Partial Response [PR], or Stable Disease [SD]), Assessed According to Response Evaluation Criteria in Solid Tumors (RECIST) and Cancer Antigen-125 (CA-125) Response Criteria (Phase II)
Time Frame: Up to 2 years
Measure: Number; unit: participants
Arm/Group | Treatment (Ixabepilone and Doxorubicin)
Number analyzed (Participants) | 45
participants
  Ovarian Cancer | 20
  Breast Cancer | 7

3. Secondary Outcome: Progression-free Survival
Description: We will summarize progression-free survival by Kaplan-Meier survival analysis.
Time Frame: The time from start of treatment to time of progression or death, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ixabepilone and Doxorubicin)
Number analyzed (Participants) | 45
months | 4.1 [2.7 to 8.2]

4. Primary Outcome: Maximum Tolerated Dose
Description: The phase I component of the study included 30 patients with breast and ovarian cancer. A protocol amendment was made during phase I trial from a treatment regimen of Schedule A (ixabepilone every 3-4 weeks) to Schedule B (ixabepilone every week). The maximum tolerated dose was determined to be the preceding dose of any dose that resulted in 2 DLT events. Schedule B was carried forward to the phase II trial. The Maximum Tolerated Dose for Schedule B is reported. Please see (Chuang et al., 2010) for additional details
Time Frame: Once 2 DLT events occur in patients during the first 28 days of treatment (cycle 1), the preceding dose will be designated the maximum tolerated dose (MTD).
Population: The phase I component of the study included 30 patients with breast and ovarian cancer.
Measure: Number; unit: mg/m2
Arm/Group | Treatment (Ixabepilone and Doxorubicin)
Number analyzed (Participants) | 30
mg/m2 | 16

ADVERSE EVENTS:
Groups:
- Ixabepilone 24mg/m2 and Doxorubicin 30mg/m2: Level 1; Ixabepilone 32mg/m2 and Doxorubicin 30mg/m2: Level 2; Ixabepilone 40mg/m2 and Doxorubicin 30mg/m2: Level 3: Ixabepilone IV over 3 hours and pegylated liposomal doxorubicin hydrochloride IV over 30-60 minutes on day 1.
  ixabepilone: Given IV
  pegylated liposomal doxorubicin hydrochloride: Given IV
- Ixabepilone 13mg/m2 and Doxorubicin 30mg/m2: Level 4; Ixabepilone 16mg/m2 and Doxorubicin 30mg/m2: Level 5: Ixabepilone IV over 3 hours on days 1, 8 and 15 and pegylated liposomal doxorubicin hydrochloride IV over 30-60 minutes on day 1
  ixabepilone: Given IV
  pegylated liposomal doxorubicin hydrochloride: Given IV
Arm/Group | Ixabepilone 24mg/m2 and Doxorubicin 30mg/m2: Level 1 | Ixabepilone 32mg/m2 and Doxorubicin 30mg/m2: Level 2 | Ixabepilone 40mg/m2 and Doxorubicin 30mg/m2: Level 3 | Ixabepilone 13mg/m2 and Doxorubicin 30mg/m2: Level 4 | Ixabepilone 16mg/m2 and Doxorubicin 30mg/m2: Level 5
Serious Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 3/3 | 24/24
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 3/3 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixabepilone 24mg/m2 and Doxorubicin 30mg/m2: Level 1 (N=6) | Ixabepilone 32mg/m2 and Doxorubicin 30mg/m2: Level 2 (N=6) | Ixabepilone 40mg/m2 and Doxorubicin 30mg/m2: Level 3 (N=6) | Ixabepilone 13mg/m2 and Doxorubicin 30mg/m2: Level 4 (N=3) | Ixabepilone 16mg/m2 and Doxorubicin 30mg/m2: Level 5 (N=24)
Blood Bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CNS cerebrovascular ischemia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Hemorrhage, pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with grade 3 or 4 neutrophils (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Neuropathy: Sensory (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophils count decreased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 5 (5)
Rash: desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Lung infections (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death NOS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixabepilone 24mg/m2 and Doxorubicin 30mg/m2: Level 1 (N=6) | Ixabepilone 32mg/m2 and Doxorubicin 30mg/m2: Level 2 (N=6) | Ixabepilone 40mg/m2 and Doxorubicin 30mg/m2: Level 3 (N=6) | Ixabepilone 13mg/m2 and Doxorubicin 30mg/m2: Level 4 (N=3) | Ixabepilone 16mg/m2 and Doxorubicin 30mg/m2: Level 5 (N=24)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2) | 2 (2) | 11 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 4 (4)
Anorexia (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 7 (7)
Rash maculo-papular (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 6 (6)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 6 (6)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Fatigue (General disorders) | 3 (3) | 3 (3) | 0 (0) | 3 (3) | 15 (15)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 6 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 6 (6)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 10 (10)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 6 (6)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 7 (7)
Vaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 7 (7)
Hand and foot syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 9 (9)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (5)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
skin infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 5 (5)
Dehydration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic Pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rash: acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less